CLINICAL TRIAL: NCT03856502
Title: Impact of Intrathecal Dexamethasone Administration for Elderly Patients With Proximal Femoral Fracture
Brief Title: Influence of Intrathecal Dexamethasone Administration for Proximal Femoral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital Sveti Duh (Other)
Responsible Party: Principal Investigator, Livija Šakić, MD,PhD, MD,PhD Anesthesiology, Reanimatology and Intensive Medicine, General Hospital Sveti Duh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 662809198348
Record Dates: First submitted 2018-11-02; First posted 2019-02-27 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Femoral Fracture; Cognition Disorders; Cortisol; Hypersecretion
Keywords: spinal anesthesia; femoral fracture; dexamethasone
MeSH Terms: conditions — Femoral Fractures; Cognition Disorders | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- group that received dexamethasone (DLSA) (Experimental): The study group of 30 patients ASA status 2 or 3 received 8 mg of dexamethasone with 12,5 mg of 0,5% of levobupivacaine intrathecally for surgical reconstruction of proximal femoral fracture. Spinal anaesthesia was performed in sitting position using middle approach in intervertebral space L2-L3 or L3-L4 with spinal needles 22-27 GA.
  Interventions: Drug: 8 mg of dexamethasone; Drug: 12,5 mg of 0,5 % of levobupivacaine
- group without dexamethasone (LSA) (Active Comparator): The control group of 30 patients ASA status 2 or 3 received 12,5 mg of 0,5% of levobupivacaine intrathecally for surgical reconstruction of proximal femoral fracture. Spinal anaesthesia was performed in sitting position using middle approach in intervertebral space L2-L3 or L3-L4 with spinal needles 22-27 GA.
  Interventions: Drug: 12,5 mg of 0,5 % of levobupivacaine

INTERVENTIONS:
Drug: 8 mg of dexamethasone — Effect of intrathecally administered dexamethasone in spinal anaesthesia for surgical correction of the hip fracture.
  Other Names: Dexamethasone KRKA, Chirocaine Abbott
  Arms: group that received dexamethasone (DLSA)
Drug: 12,5 mg of 0,5 % of levobupivacaine — Local anaesthetic standardly used in spinal anaesthesia for surgical correction of the hip fracture by the particular hospital's protocol.
  Other Names: Chirocaine Abbott

SUMMARY:
Spinal anesthesia blocks acute pain in older patients with femur fracture. Delirium is a common complication seen after femur fracture, affecting approximately 10-16% of patients. It is associated with increased mortality at 1st year, delayed rehabilitation efforts, prolonged length of hospital stay, poorer functional outcomes, and increased risk of nursing home placement.

Intrathecal dexamethasone administration improves quality of anesthesia in patients with femur fracture compared to conventional spinal anesthesia.

DETAILED DESCRIPTION:
The aim of this research was to establish the influence of intrathecal dexamethasone administration in spinal anaesthesia with levobupivacaine on postoperative pain and changes of consciousness, values of cortisol levels and quality of treatment for patients with femoral fractures compared to spinal anaesthesia with only local anaesthetic.

The study was planned as a prospective, observational, randomised clinical trial. A total of 60 patients ASA2 and ASA3 status, scheduled for surgical procedures were sorted into two groups and underwent surgery in spinal anesthesia with levobupivacaine with or without dexamethsone.

ELIGIBILITY:
Inclusion Criteria:

* cooperative ASA 2 and ASA 3 status patients with proximal femoral fractures of one leg
* agreed to be enrolled in the study (Informed Consent signed)

Exclusion Criteria:

* patients refused to be enrolled in the study
* patients with pre-existing cognitive disturbances before surgery
* conditions or diseases with corticosteroid therapy, long term corticosteroid, diabetes mellitus, neurological conditions or tumors, neuroendocrine disorders or tumors
* breaking the study protocols
* patients who no longer wanted to be enrolled in the study
* unexpected events when the study already started

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11-11 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
postoperative cognitive change | Confusion Assessment Method scoring was assessed in 4 measure points: 1. one hour after surgery, 2. on the 3rd postoperative day at 9 am, 3. on the 5th postoperative day at 9 am, 4. on the 10th postoperative day at 9 am
  Assessed using a simplified Confusion Assessment Method scoring scale, a clinical instrument for delirium assessment used by non-psychiatric medical staff after surgery for excluding delirium. Delirium is defined in terms of 4 possible diagnostic criteria (1. acute onset or fluctuating course; 2- inattention; 3- disorganised thinking; 4- altered level of consciousness (may be defined as alert, lethargic, stupor or coma cognitive state)) and is defined as present when 1 plus 2 and either 3 or 4 diagnostic criteria are positive.
cortisol concentrations changes | Measured in 5 measure points: 1. one hour before surgery, 2. one hour after surgery, 3. on the 3rd postoperative day at 6 am, 4. on the 5th postoperative day at 6 am, 5. on the 10th postoperative day at 6 am
  Determined from patient's blood plasma assessed by Roche Elecsys Immunoassay System and defined from the laboratory reference points (185-624)nmol/L equal for each measure point; for single measuring 0,5 ml of patient's blood was taken

SECONDARY OUTCOMES:
perioperative pain intensity: Visual Analogue Scale score | Visual Analogue Scale scoring (scores: 0-10) was assessed in 5 measure points every 3 hours when patient was awake: 1. 1 h before surgery, 2. 1 h after surgery, 3. on the 3rd postoperative day, 4. on the 5th postoperative day, 5. 10th postoperative day
  Assessed using Visual Analogue Scale score and establishing postoperative analgesic requirements
glucose concentrations changes | Measured in 5 measure points (units: mmol/L): 1. one hour before surgery, 2. one hour after surgery, 3. on the 3rd postoperative day at 6 am, 4. on the 5th postoperative day at 6 am, 5. on the 10th postoperative day at 6 am
  Determined form patient's blood plasma assessed by Beckman Coulter AU400 and AU680 orbOlympus Glucose Analyzer 2 devices defined from the laboratory reference points (4,4-6,4)mmol/L equal for each measure point; for single measuring 0,2 ml of patient's blood was taken
Blood loss | During the surgical repairment and up to the removal of drainage systems (2nd postoperative day)
  Determinated by intraoperative blood loss in mililitres, amount of blood in drainage systems in mililitres, transfusion of homologous blood in mililitres
Number of Participants with pulmonary embolism | During surgical reconstruction and during postoperative follow-up of up to ten postoperative days
  Established by noted pulmonary embolism in the operating room or at the traumatology ward by the ward staff
Number of Participants with heart failure | During surgical reconstruction and during postoperative follow-up of up to ten postoperative days
  Established by noted heart failure in the operating room or at the traumatology ward by the ward staff
Platelets changes | Assessed in 5 measure points: 1.one hour before surgery, 2. one hour after surgery, 3. on the 3rd postoperative day at 6 am, 4. on the 5th postoperative day at 6 am, 5. on the 10th postoperative day at 6 am
  Determined from laboratory values of platelets data in reference points (158-424)10^9/L equal for each measure point
Haemoglobin changes | Assessed in 5 measure points: 1.one hour before surgery, 2. one hour after surgery, 3. on the 3rd postoperative day at 6 am, 4. on the 5th postoperative day at 6 am, 5. on the 10th postoperative day at 6 am
  Determined from laboratory values of haemoglobin data measured reference points (119-157)g/L equal for each measure point
Haematocrit changes | Assessed in 5 measure points: 1.one hour before surgery, 2. one hour after surgery, 3. on the 3rd postoperative day at 6 am, 4. on the 5th postoperative day at 6 am, 5. on the 10th postoperative day at 6 am
  Determined from laboratory values of haematocrit data in reference points (0,356-0,470)L/L equal for each measure point
Hospitalisation | In the time period of up to 30 days
  Calculated by number of days preoperatively from the day of admission to the day of surgical treatment and postoperatively from the day of surgical treatment to the day of hospital discharge
Number of Participants who underwent surgical procedure during first 48 hours from admission | Calculated in hours after the patient's admission to the hospital's Emergency Department to the point of surgical reconstruction in the time period up to 48 hours
  It was defined if surgical procedure was performed in first 48 hours from admission to the hospital's Emergency Department or later reflecting morbidity and/or mortality

CONTACTS AND LOCATIONS:
Overall Officials: Livija Šakić, MD,PhD, Principal Investigator — University Hospital Sveti Duh
Locations (1):
- University Hospital "Sveti Duh", Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No
The research has been a doctoral thesis.

REFERENCES:
- [Background] Neuman MD, Silber JH, Elkassabany NM, Ludwig JM, Fleisher LA. Comparative effectiveness of regional versus general anesthesia for hip fracture surgery in adults. Anesthesiology. 2012 Jul;117(1):72-92. doi: 10.1097/ALN.0b013e3182545e7c. PMID 22713634
- [Background] Membership of the Working Party; Griffiths R, Alper J, Beckingsale A, Goldhill D, Heyburn G, Holloway J, Leaper E, Parker M, Ridgway S, White S, Wiese M, Wilson I. Management of proximal femoral fractures 2011: Association of Anaesthetists of Great Britain and Ireland. Anaesthesia. 2012 Jan;67(1):85-98. doi: 10.1111/j.1365-2044.2011.06957.x. PMID 22150501
- [Background] Borgeat A, Ekatodramis G. Orthopaedic surgery in the elderly. Best Pract Res Clin Anaesthesiol. 2003 Jun;17(2):235-44. doi: 10.1016/s1521-6896(03)00007-7. PMID 12817917
- [Background] Baumann H, Gauldie J. The acute phase response. Immunol Today. 1994 Feb;15(2):74-80. doi: 10.1016/0167-5699(94)90137-6. PMID 7512342
- [Background] Buckingham JC. Stress and the hypothalamo-pituitary-immune axis. Int J Tissue React. 1998;20(1):23-34. No abstract available. PMID 9561443
- [Background] Munck A, Guyre PM, Holbrook NJ. Physiological functions of glucocorticoids in stress and their relation to pharmacological actions. Endocr Rev. 1984 Winter;5(1):25-44. doi: 10.1210/edrv-5-1-25. PMID 6368214
- [Background] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999
- [Background] Hogevold HE, Lyberg T, Kahler H, Haug E, Reikeras O. Changes in plasma IL-1beta, TNF-alpha and IL-6 after total hip replacement surgery in general or regional anaesthesia. Cytokine. 2000 Jul;12(7):1156-9. doi: 10.1006/cyto.2000.0675. PMID 10880268
- [Background] Kehlet H. Manipulation of the metabolic response in clinical practice. World J Surg. 2000 Jun;24(6):690-5. doi: 10.1007/s002689910111. PMID 10773121
- [Background] Bani-Hashem N, Hassan-Nasab B, Pour EA, Maleh PA, Nabavi A, Jabbari A. Addition of intrathecal Dexamethasone to Bupivacaine for spinal anesthesia in orthopedic surgery. Saudi J Anaesth. 2011 Oct;5(4):382-6. doi: 10.4103/1658-354X.87267. PMID 22144925
- [Background] Kroin JS, Schaefer RB, Penn RD. Chronic intrathecal administration of dexamethasone sodium phosphate: pharmacokinetics and neurotoxicity in an animal model. Neurosurgery. 2000 Jan;46(1):178-82; discussion 182-3. PMID 10626948
- [Background] Yao XL, Cowan MJ, Gladwin MT, Lawrence MM, Angus CW, Shelhamer JH. Dexamethasone alters arachidonate release from human epithelial cells by induction of p11 protein synthesis and inhibition of phospholipase A2 activity. J Biol Chem. 1999 Jun 11;274(24):17202-8. doi: 10.1074/jbc.274.24.17202. PMID 10358078
- [Background] Dong Y, Zhang X, Tang F, Tian X, Zhao Y, Zhang F. Intrathecal injection with methotrexate plus dexamethasone in the treatment of central nervous system involvement in systemic lupus erythematosus. Chin Med J (Engl). 2001 Jul;114(7):764-6. PMID 11780346
- [Background] Williams BA, Hough KA, Tsui BY, Ibinson JW, Gold MS, Gebhart GF. Neurotoxicity of adjuvants used in perineural anesthesia and analgesia in comparison with ropivacaine. Reg Anesth Pain Med. 2011 May-Jun;36(3):225-30. doi: 10.1097/AAP.0b013e3182176f70. PMID 21519308
- [Background] Benzon HT, Chew TL, McCarthy RJ, Benzon HA, Walega DR. Comparison of the particle sizes of different steroids and the effect of dilution: a review of the relative neurotoxicities of the steroids. Anesthesiology. 2007 Feb;106(2):331-8. doi: 10.1097/00000542-200702000-00022. PMID 17264728
- [Background] Kopacz DJ, Lacouture PG, Wu D, Nandy P, Swanton R, Landau C. The dose response and effects of dexamethasone on bupivacaine microcapsules for intercostal blockade (T9 to T11) in healthy volunteers. Anesth Analg. 2003 Feb;96(2):576-82, table of contents. doi: 10.1097/00000539-200302000-00050. PMID 12538215
- [Background] Macro M, Reznik Y, Leymarie P, Loyau G, Mahoudeau J. The effect of intrathecal dexamethasone injection on plasma cortisol level. Br J Rheumatol. 1991 Jun;30(3):238. doi: 10.1093/rheumatology/30.3.238. No abstract available. PMID 2049597
- [Background] Bjorkelund KB, Hommel A, Thorngren KG, Gustafson L, Larsson S, Lundberg D. Reducing delirium in elderly patients with hip fracture: a multi-factorial intervention study. Acta Anaesthesiol Scand. 2010 Jul;54(6):678-88. doi: 10.1111/j.1399-6576.2010.02232.x. Epub 2010 Mar 15. PMID 20236093
- [Background] Rasmussen LS, O'Brien JT, Silverstein JH, Johnson TW, Siersma VD, Canet J, Jolles J, Hanning CD, Kuipers HM, Abildstrom H, Papaioannou A, Raeder J, Yli-Hankala A, Sneyd JR, Munoz L, Moller JT; ISPOCD2 Investigators. Is peri-operative cortisol secretion related to post-operative cognitive dysfunction? Acta Anaesthesiol Scand. 2005 Oct;49(9):1225-31. doi: 10.1111/j.1399-6576.2005.00791.x. PMID 16146456
- [Background] Mouzopoulos G, Vasiliadis G, Lasanianos N, Nikolaras G, Morakis E, Kaminaris M. Fascia iliaca block prophylaxis for hip fracture patients at risk for delirium: a randomized placebo-controlled study. J Orthop Traumatol. 2009 Sep;10(3):127-33. doi: 10.1007/s10195-009-0062-6. Epub 2009 Aug 19. PMID 19690943
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Huang YF, Liang J, Shyu YL. Number of Comorbidities Negatively Influence Psychological Outcomes of the Elderly Following Hip Fracture in Taiwan. J Aging Health. 2016 Dec;28(8):1343-1361. doi: 10.1177/0898264315618922. Epub 2016 Jul 8. PMID 26786859
- [Background] Drews T, Franck M, Radtke FM, Weiss B, Krampe H, Brockhaus WR, Winterer G, Spies CD. Postoperative delirium is an independent risk factor for posttraumatic stress disorder in the elderly patient: a prospective observational study. Eur J Anaesthesiol. 2015 Mar;32(3):147-51. doi: 10.1097/EJA.0000000000000107. PMID 24979586
- [Background] Le Manach Y, Collins G, Bhandari M, Bessissow A, Boddaert J, Khiami F, Chaudhry H, De Beer J, Riou B, Landais P, Winemaker M, Boudemaghe T, Devereaux PJ. Outcomes After Hip Fracture Surgery Compared With Elective Total Hip Replacement. JAMA. 2015 Sep 15;314(11):1159-66. doi: 10.1001/jama.2015.10842. PMID 26372585
- Available data/document: Individual Participant Data Set — https://hrcak.srce.hr/106014
- Available data/document: Individual Participant Data Set — https://hrcak.srce.hr/143046
- Available data/document: Individual Participant Data Set — https://www.bib.irb.hr/889771
- Available data/document: Individual Participant Data Set — https://www.bib.irb.hr/889781
- Available data/document: Individual Participant Data Set — https://www.bib.irb.hr/889773